CLINICAL TRIAL: NCT02792413
Title: Randomized Controlled Study Evaluating the Effect of a Biotherapy Treatment (Anti-RANKL Ligand Antibody: Denosumab) on Bone and Vascular Metabolism in Osteoporotic Chronic Kidney Disease
Brief Title: Study Evaluating Denosumab on Bone and Vascular Metabolism in Osteoporotic Chronic Kidney Disease
Acronym: HDENO
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Modified study and new deposit in RECHMPL21_0451
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RECHMPL15_0496; UF 9676 (Other: Montpellier University Hospital)
Record Dates: First submitted 2016-06-02; First posted 2016-06-07 (Estimated); Last update posted 2023-08-09 (Actual); Status verified 2022-04

CONDITIONS: Female With Osteoporosis and Chronic Kidney Disease
Keywords: osteoporosis; chronic kidney disease; anti-RANK ligand antibody; bone mineral density; vascular calcifications
MeSH Terms: conditions — Renal Insufficiency, Chronic; Osteoporosis; Vascular Calcification | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Denosumab (Experimental): Denosumab 60 mg, subcutaneous injection every 6 months for 24 months
  Interventions: Drug: Denosumab
- Placebo (Placebo Comparator): NaCl 0.9% (1 mL), subcutaneous injection every 6 months for 24 months
  Interventions: Drug: NaCl (placebo)

INTERVENTIONS:
Drug: Denosumab — Patients will receive a subcutaneous injection of Denosumab every 6 months for the duration of the study. In addition, they will receive vitamin D and calcium (which is the normal treatment) for the duration of the study.
  Arms: Denosumab
Drug: NaCl (placebo) — Patients will receive a subcutaneous injection of NaCl every 6 months for the duration of the study. In addition, they will receive vitamin D and calcium (which is the normal treatment) for the duration of the study.
  Arms: Placebo

SUMMARY:
Aim of this study is to evaluate in a population of old osteoporotic chronic kidney disease females the effect of denosumab:

* on bone mineral density (femoral T-score) at 24 months
* on bone mineral density evolution (femoral T-score) after 24 months of follow-up
* on bone mineral density evolution (lumbar T-score) after 24 months of follow-up
* on coronary and abdominal aorta calcification scores evolution after 24 months of follow-up
* on parameters of bone remodelling (OPG, RANKL, sclerostin, DKK-1), of mineral and calcium metabolism (FGF23 Ct, Klotho, PTH, 25(OH) vitamin D3, phosphorus, calcium, bone alklaline phosphatase, osteocalcin, CTX), of inflammation (CRP) after 24 months of follow-up
* on cardiovascular morbidity (cardiovascular events) and mortality after 24 months of follow-up
* the tolerance after 24 months of follow-up

DETAILED DESCRIPTION:
Aim of this study is to evaluate in a population of old osteoporotic chronic kidney disease females the effect of denosumab:

* on bone mineral density (femoral T-score) (by bone densitometry) at 24 months
* on bone mineral density evolution (femoral T-score) (by bone densitometry) after 24 months of follow-up
* on bone mineral density evolution (lumbar T-score) (by bone densitometry) after 24 months of follow-up
* on coronary and abdominal aorta calcification scores evolution (by multiple detector computed tomography and plain abdominal X-ray) after 24 months of follow-up
* on parameters of bone remodelling (OPG, RANKL, sclerostin, DKK-1), of mineral and calcium metabolism (FGF23 Ct, Klotho, PTH, 25(OH) vitamin D3, phosphorus, calcium, bone alklaline phosphatase, osteocalcin, CTX), of inflammation (CRP) after 24 months of follow-up
* on cardiovascular morbidity (cardiovascular events) and mortality after 24 months of follow-up
* the tolerance after 24 months of follow-up

ELIGIBILITY:
Inclusion Criteria:

* Patient of 65 years or older
* Chronic kidney disease stage 5 patient, hemodialyzed with extracorporeal treatment for at least 3 months
* Patient with osteoporosis (history of bone fracture or T-scoring < -2.5 SD)
* PTH levels in the serum in agreement with the KDIGO guidelines, in the absence of treatment with Cinacalcet.

Exclusion Criteria:

* Cinacalcet treatment
* Calcium parameters (PTH, 25(OH) vitamin D3, Calcium) outside the KDIGO guidelines
* Suspicion of lower bone remodeling
* Hypersensibility to active substance or one of excipients of denosumab
* Patient with a cancer or myeloma
* Patient with severe heaptic cytolysis
* Patients with severe teeth problems
* Patient positive for HIV
* Patient involved in another biomedical research
* Vulnerable patients (protected by the law, under guardianship, deprived of freedom)

Ages: 65 Years to 95 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Relative variation of femoral bone mineral density after 24 months of follow-up (T-score evaluated by osteodensitometry) | 24 months after inclusion

SECONDARY OUTCOMES:
Relative variation of lumbar bone mineral density after 24 months of follow-up (T-score evaluated by osteodensitometry) | 24 months after inclusion
Relative variation of coronary calcification scores after 24 months of follow-up | 24 months after inclusion
Relative variation of abdominal aorta calcification scores after 24 months of follow-up | 24 months after inclusion
Variation of calcium at 6, 12, 18 and 24 months of follow-up | 6, 12, 18 and 24 months after inclusion
Variation of phosphorus at 6, 12, 18 et 24 months of follow-up | 6, 12, 18 and 24 months after inclusion
Morbi-mortality at 24 months of follow-up | 24 months after inclusion
Adverse events occuring during the entire study | 24 months after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul CRISTOL, Prof, Principal Investigator — CHU Lapeyronie, Department of Biochemistry and Hormonology, Montpellier, FRANCE
Locations (9):
- France (9):
  - Clinique Médipole Cabestany, Cabestany
  - CHL Castelnau Le Lez, Castelnau-le-Lez
  - CHU Lyon Sud, Nephrology department, Lyon
  - AP-HM, Nephrology department, Marseille
  - AIDER, Montpellier
  - CHU Montpellier, Nephrology department, Montpellier
  - CHU Nice, Nephrology department, Nice
  - CHU Nimes, Nephrology department, Nîmes
  - CH Perpignan, Nephrology department, Perpignan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hara T, Hijikata Y, Matsubara Y, Watanabe N. Pharmacological interventions versus placebo, no treatment or usual care for osteoporosis in people with chronic kidney disease stages 3-5D. Cochrane Database Syst Rev. 2021 Jul 7;7(7):CD013424. doi: 10.1002/14651858.CD013424.pub2. PMID 34231877